CLINICAL TRIAL: NCT01897701
Title: A Phase 1 Randomized, Observer-Blinded, Dose-Ranging Study to Evaluate the Immunogenicity and Safety of Monovalent A/Anhui/1/2013 (H7N9) Virus-Like Particle (VLP) Avian Influenza Antigen (Recombinant) in Healthy Adults With and Without Adjuvant 1
Brief Title: A(H7N9) VLP Antigen Dose Ranging Study With Adjuvant 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NVX900.PH7.101
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Avian Influenza
Keywords: H7N9
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Group A (Experimental): High dose Monovalent Avian Influenza VLP (H7N9); IM; Day 0 & 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9)
- Group B (Experimental): Intermediate dose Monovalent Avian Influenza VLP (H7N9); IM; Day 0 & 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9)
- Group C (Experimental): Intermediate dose Monovalent Avian Influenza VLP (H7N9) and Low dose Adjuvant 1; IM; Day 0 & 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9); Biological: Adjuvant 1
- Group D (Experimental): Low dose Monovalent Avian Influenza VLP (H7N9) and Low dose Adjuvant 1; IM; Day 0 & Day 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9); Biological: Adjuvant 1
- Group E (Experimental): Intermediate dose Monovalent Avian Influenza VLP (H7N9) and High dose Adjuvant 1; IM; Day 0 & 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9); Biological: Adjuvant 1
- Group F (Experimental): Low dose Monovalent Avian Influenza VLP (H7N9) and High dose Adjuvant 1; IM; Day 0 & 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9); Biological: Adjuvant 1
- Group G (Experimental): Placebo; IM; Day 0 & 21
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Monovalent Avian Influenza VLP (H7N9)
  Arms: Group A; Group B; Group C; Group D; Group E; Group F
Biological: Adjuvant 1
  Arms: Group C; Group D; Group E; Group F
Biological: Placebo
  Arms: Group G

SUMMARY:
This is a randomized, observer-blinded, placebo-controlled trial in adults ≥18 years old. Randomization will be stratified by age (18 to 49 years and ≥50 years) and by prior influenza immunization within the past three months. Proportions of subjects in the various strata will not be pre-specified; rather, the goal will be to achieve an approximately equal distribution of subjects with these characteristics across the various treatment groups.

Treatments will comprise two identical IM doses at a 21-day interval (Day 0 and Day 21), in alternate deltoids. For each subject, study follow-up will span approximately 385 days total, or approximately 13 months from the first dose.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following to be eligible for participation in the study:

1. Healthy adult male or female, ≥18 years of age,
2. Willing and able to give informed consent prior to study enrollment,
3. Able to comply with study requirements, and
4. Women of childbearing potential must have a negative urine pregnancy test prior to each vaccination, will be advised through the Informed Consent process to avoid becoming pregnant over the duration of the study, and must assert that they will employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: credible history of continuous abstinence from heterosexual activity or prior surgical sterilization, hormonal contraceptives (oral, injectable, implant, patch, ring), barrier contraceptives (condom or diaphragm), and intrauterine device (IUD). Women with an adequately documented history of surgical sterility, or ≥50 years of age and without menses for ≥ 1 year are exempt from urine pregnancy testing.

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for participation in the study.

1. Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care.

   * Asymptomatic conditions or findings (e.g., mild hypertension, dyslipidemia) that are not associated with evidence of end-organ damage are not exclusionary provided that they are being appropriately managed and are clinically stable (i.e., unlikely to result in symptomatic illness within the time-course of this study) in the opinion of the investigator.
   * Note that illnesses or conditions may be exclusionary, even if otherwise stable, due to therapies used to treat them (see exclusion criteria 2, 5, 7, 8).
2. Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of first vaccination.
3. History of a serious reaction to prior influenza vaccination.
4. History of Guillain-Barré Syndrome (GBS) within 6 weeks following a previous influenza vaccine.
5. Received any vaccine in the 4 weeks preceding the study vaccination; or any A(H7N9) avian influenza vaccine at any time.
6. Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
7. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
8. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
9. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C on the planned day of vaccine administration).
10. Known disturbance of coagulation.
11. Women who are pregnant or breastfeeding, or plan to become pregnant during the study.
12. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.
13. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
14. Persons employed in a capacity that involves handling poultry or wild birds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Assessment of Safety | Day 0 to Day 384
  Number (and percentages) of subjects with solicited local and systemic AEs over the seven days post-injection and all adverse events, solicited and unsolicited, including adverse changes in clinical laboratory parameters, over 35 days post-first injection.
  Significant New Medical Conditions, Medically Attended Events and Serious Adverse Events will be collected for one year post-second injection.
Immunogenicity as assessed by hemagglutination-inhibiting (HAI) antibody titers against the vaccine-homologous A/Anhui/1/13 (H7N9) virus. | Day 0 to Day 384
  * Geometric mean titer (GMT)
  * Geometric mean ratio (GMR)
  * Seroconversion rate (SCR)
  * Seroresponse rate (SRR)

SECONDARY OUTCOMES:
Immunogenicity as assessed by neuraminidase-inhibiting antibodies to N9. | Day 0 to Day 384

CONTACTS AND LOCATIONS:
Overall Officials: D. Nigel Thomas, Ph.D., Study Director — Novavax, Inc.
Locations (3):
- Australia (3):
  - Q-Pharm Pty Limited, Herston, Queensland
  - CMAX, Adelaide, South Australia
  - Linear Clinical Research, Nedlands, Western Australia

REFERENCES:
- [Derived] Fries LF, Smith GE, Glenn GM. A recombinant viruslike particle influenza A (H7N9) vaccine. N Engl J Med. 2013 Dec 26;369(26):2564-6. doi: 10.1056/NEJMc1313186. Epub 2013 Nov 13. No abstract available. PMID 24224560
- See also: Novavax Homepage — http://novavax.com/